CLINICAL TRIAL: NCT01140542
Title: Efficacy of 500µg Roflumilast Once Daily Versus Placebo Over 12 Weeks in Patients With Diabetes Mellitus Type 2. A Double Blind, Parallel Group, Phase IIb, Proof of Concept Clinical Study
Brief Title: Efficacy of 500µg Roflumilast Once Daily Versus Placebo Over 12 Weeks in Patients With Diabetes Mellitus Type 2. A Double Blind, Parallel Group, Proof of Concept Clinical Study
Acronym: FORTUNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY217/M2-401
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-09

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes Mellitus Type 2; Roflumilast
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Roflumilast (Active Comparator): 500µg, once daily
  Interventions: Drug: Roflumilast
- Placebo (Placebo Comparator)
  Interventions: Drug: Roflumilast

INTERVENTIONS:
Drug: Roflumilast — 500µg, once daily

SUMMARY:
This study is a proof of concept study to confirm in a standardized manner the therapeutic efficacy of roflumilast in type 2 diabetes mellitus patients.

ELIGIBILITY:
Inclusion Criteria:

* given written informed consent
* patients with diagnosis of type 2 diabetes according to American Diabetes Association (ADA) criteria and inadequately controlled on diet and exercise alone
* HbA1c at baseline: ≥7.5 percent to 8.5 percent (up to 9 percent in Mexico, Ukraine and Romania)
* BMI between ≥26 and ≤35 kg/m2
* willingness of patient to check his/her blood glucose with equipment provided by the sponsor during the treatment phase in case of hypo-/hyperglycemia episodes
* willingness to adhere to the physician's advise to comply with diet and exercise

Main Exclusion Criteria:

* patients diagnosed with type 1 diabetes or diabetes secondary to pancreatitis or resection of pancreas
* patients diagnosed with hemoglobinopathies, hemolytic anemia or other diseases which interfere with HbA1c measurement
* non-euthyroid patients or patients with a non-controlled hypo- or hyperthyroidism
* reported gain or loss of more than 5 percent of body weight within the last 2 months prior to V0
* treatment with any diabetes medication prior to V0
* treatment with any weight-loss medication within 3 months prior to V0
* treatment with any not allowed medication or nutrition additives
* clinically relevant abnormal laboratory values suggesting an unknown disease and requiring further clinical evaluation (as assessed by the investigator)
* clinically significant cardiac abnormalities (diagnosed clinically, or by X-ray/ECG) that were not related to type 2 diabetes mellitus and that required further evaluation
* participation in a clinical study with study medication for weight loss or type 2 diabetes

Patients were randomized after 2 weeks of the baseline period, if the following criteria were fulfilled:

* judged to be clinically stable
* tablet compliance ≥80 percent and ≤125 percent
* HbA1c in the range of 7.5 percent to 8.5 percent (up to 9 percent in Mexico, Ukraine and Romania) tested at V0 by the central laboratory

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2006-08; Primary Completion 2007-11 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c [percent] from baseline to the last study visit (Vlast) | Baseline to last visit

SECONDARY OUTCOMES:
Mean change in HbA1c from baseline to each scheduled post-randomization visit
Mean change from baseline to each scheduled post-randomization visit and Vlast in blood parameters
  blood parameters: serum lipids (high-density-lipoprotein-cholesterol [HDL], low-density-lipoprotein-cholesterol [LDL], and triglycerides [TG]), fasting plasma glucose (FPG), fructosamine, glycerol, free fatty acids [FFA], plasma insulin, fasting pro-insulin, cholesterol, c-reactive protein (CRP), interleukin-6 (IL-6), TNF-α, intercellular adhesion molecule 1 (ICAM-1), E-selectin, plasminogen activator inhibitor 1 (PAI-1), adiponectin, and leptin
Mean change from baseline to each scheduled post-randomization visit and Vlast based on a 5-hour period post meal area under the curve (AUC) for FFA, glycerol, glucose, glucagons, insulin, and C-peptide
Mean change in body weight, waist and hip circumference, waist to hip ratio, and body mass index (BMI) from baseline to each scheduled post-randomization visit and Vlast
Time to event (study withdrawal, time to study withdrawal due to an adverse event (AE) and time to lack of efficacy (LOE)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca

REFERENCES:
- See also: BY217-M2-401-RDS-2009-01-14-.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4496&filename=BY217-M2-401-RDS-2009-01-14-.pdf